CLINICAL TRIAL: NCT03023124
Title: Solitary Fibrous Tumor: Phase II Study on Trabectedin Versus Adriamycin Plus Dacarbazine in Advanced Patients
Brief Title: Study With Trabectedin Versus Adriamycin Plus Dacarbazine, in Patients With Advanced Solitary Fibrous Tumor
Acronym: STRADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISG STRADA
Record Dates: First submitted 2016-12-19; First posted 2017-01-18 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-02

CONDITIONS: Solitary Fibrous Tumors
MeSH Terms: conditions — Solitary Fibrous Tumors | interventions — Trabectedin; Doxorubicin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabectedin (Experimental): trabectedin: 1.5 mg/m² - 1.3 mg/m² given in 24-hour continuous infusion every 21 days for 6 cycles
  Interventions: Drug: Trabectedin
- Adriamycin and Dacarbazine (Experimental): Adriamycin: 75 mg/m2/day, bolus, day 1 every 21 days for 6 cycles Dacarbazine: 400 mg/m2/day, days 1, 2 every 21 days for 6 cycles
  Interventions: Drug: Adriamycin; Drug: Dacarbazine

INTERVENTIONS:
Drug: Trabectedin — Treatment with trabectedin repeated every 21 days for 6 cycles
  Arms: Trabectedin
Drug: Adriamycin — Treatment with Adriamycin at day 1 every 21 days for 6 cycles
  Arms: Adriamycin and Dacarbazine
Drug: Dacarbazine — Treatment with Dacarbazine at days 1 and 2 every 21 days for 6 cycles
  Arms: Adriamycin and Dacarbazine

SUMMARY:
Phase II randomized study for the comparison of trabectedin versus doxorubicin plus dacarbazine in patients with advanced solitary fibrous tumor

DETAILED DESCRIPTION:
Patients with solitary fibrous tumor will be randomized to receive 6 cycles of trabectedin or doxorubicin plus dacarbazine.

In case of progression or unacceptable toxicity while under the experimental treatment prior to the completion of the 6 cycles, the patients will be offered to cross to the other arm (trabectedin arm to doxorubicin plus dacarbazine arm and vice versa).

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legal representative must be able to read and understand the informed consent form (ICF) and must have been willing to give written informed consent and any locally required authorisation before any study-specific procedures, including screening evaluations, sampling, and analyses.
2. Age ≥18 years
3. Histological centrally and molecularly confirmed diagnosis of solitary fibrous tumor (inclusive of the last available tumor sample)
4. Locally advanced disease (i.e. surgical resection of local disease unfeasible radically, or unaccepted by the patient, or amenable to become less demolitive, or feasible, or easier, after cytoreduction) and/or metastatic disease
5. Measurable or evaluable disease with RECIST
6. Evidence of progression by RECIST during the 6 months before study entry
7. Patients must be cytotoxic chemotherapy naïve (patients treated with neoadjuvant/adjuvant chemotherapy cannot be included) or could have received a previous target agent in front-line setting.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
9. Adequate bone marrow function
10. Adequate organ function
11. Cardiac ejection fraction ≥50% as measured by echocardiogram
12. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation each cycle of chemotherapy. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study.
13. No history of arterial and/or venous thromboembolic event within the previous 12 months.

Exclusion Criteria:

1. Any prior treatment with cytotoxic chemotherapy
2. >1 line of anticancer targeted agents
3. Previous treatment with any other investigational or not investigational agents within 14 days of first day of study drug dosing
4. Previous treatment with radiation therapy within 14 days of first day of study drug dosing, or patients who have not recovered from adverse events due to agents previously administered
5. Previous radiotherapy to 25 % of the bone marrow
6. Major surgery within 4 weeks prior to study entry
7. Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged to entail a low risk of relapse
8. Pregnancy or breast feeding
9. Cardiovascular diseases resulting in a New York Heart Association Functional Status >2 (24). Medical history of a myocardial infarction < 6 months prior to initiation of study treatment
10. Medical history of arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months prior to the initiation of study treatment
11. Known history of human immunodeficiency virus infection
12. Active or chronic hepatitis B or C requiring treatment with antiviral therapy
13. Medical history of hemorrhage or a bleeding event ≥ Grade 3 (NCI-CTCAE v 4.0) within 4 weeks prior to the initiation of study treatment
14. Evidence of any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
15. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
16. Expected non-compliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Overall Tumor Response Rate | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first assessed up to 54 weeks.
  evaluate the activity of trabectedin and of adriamycin in combination with dacarbazine, according to Response Evaluation Criteria in Solid Tumor (RECIST), version 1.1

SECONDARY OUTCOMES:
Choi Response Rate | week 6, week 12, week 18, then every 12 weeks up to 54 weeks
  Percentage of patient who experienced Complete or Partial Responses after treatment according to Choi Criteria.
Overall Survival (OS) | From enrollment up to 5 years
  Time from the date of enrollment to date of death
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks
  Survival free of progressive disease evaluated from enrollment up to progression according to RECIST, or death
Clinical Benefit Rate (CBR) | week 6, week 12, week 18, then every 12 weeks up to 54 weeks
  Percentage of patients who have achieved complete response, partial response or stable disease ≥ 6 months
Response rate by RECIST after the cross over | week 18, week 24, week 30, week 36 and then every 12 weeks up to 54 weeks
  Percentage of patient who experienced Complete or Partial Responses according RECIST 1.1 after cross over
Progression Free Survival (PFS) after cross over up to progression according to RECIST, or death | From date of cross over until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks
  Survival free of progressive disease evaluated from
Safety according to Common Terminology Criteria for Adverse Events (CTCAE) | From enrollment every 3 weeks up to 54 weeks
  Safety profile of the treatment evaluated according to Common Terminology Criteria for Adverse Events version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, MD, Principal Investigator — Italian Sarcoma Group
Locations (6):
- Italy (6):
  - Nuovo Ospedale di Prato, Prato, Firenze
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - IRCCS Istituto ortopedico Rizzoli, Bologna
  - Fondazione Del Piemonte Per L'Oncologia Ircc Di Candiolo -, Candiolo
  - Ospedale Giaccone, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dagrada GP, Spagnuolo RD, Mauro V, Tamborini E, Cesana L, Gronchi A, Stacchiotti S, Pierotti MA, Negri T, Pilotti S. Solitary fibrous tumors: loss of chimeric protein expression and genomic instability mark dedifferentiation. Mod Pathol. 2015 Aug;28(8):1074-83. doi: 10.1038/modpathol.2015.70. Epub 2015 May 29. PMID 26022454
- [Background] Beadle GF, Hillcoat BL. Treatment of advanced malignant hemangiopericytoma with combination adriamycin and DTIC: a report of four cases. J Surg Oncol. 1983 Mar;22(3):167-70. doi: 10.1002/jso.2930220306. PMID 6682161
- [Background] Stacchiotti S, Libertini M, Negri T, Palassini E, Gronchi A, Fatigoni S, Poletti P, Vincenzi B, Dei Tos AP, Mariani L, Pilotti S, Casali PG. Response to chemotherapy of solitary fibrous tumour: a retrospective study. Eur J Cancer. 2013 Jul;49(10):2376-83. doi: 10.1016/j.ejca.2013.03.017. Epub 2013 Apr 6. PMID 23566418
- [Background] Stacchiotti S, Tortoreto M, Bozzi F, Tamborini E, Morosi C, Messina A, Libertini M, Palassini E, Cominetti D, Negri T, Gronchi A, Pilotti S, Zaffaroni N, Casali PG. Dacarbazine in solitary fibrous tumor: a case series analysis and preclinical evidence vis-a-vis temozolomide and antiangiogenics. Clin Cancer Res. 2013 Sep 15;19(18):5192-201. doi: 10.1158/1078-0432.CCR-13-0776. Epub 2013 Jul 25. PMID 23888069
- [Background] Park MS, Ravi V, Conley A, Patel SR, Trent JC, Lev DC, Lazar AJ, Wang WL, Benjamin RS, Araujo DM. The role of chemotherapy in advanced solitary fibrous tumors: a retrospective analysis. Clin Sarcoma Res. 2013 May 11;3(1):7. doi: 10.1186/2045-3329-3-7. PMID 23663788
- [Background] Chaigneau L, Kalbacher E, Thiery-Vuillemin A, Fagnoni-Legat C, Isambert N, Aherfi L, Pauchot J, Delroeux D, Servagi-Vernat S, Mansi L, Pivot X. Efficacy of trabectedin in metastatic solitary fibrous tumor. Rare Tumors. 2011 Jul 11;3(3):e29. doi: 10.4081/rt.2011.e29. Epub 2011 Jul 18. PMID 22066036
- [Background] Khalifa J, Ouali M, Chaltiel L, Le Guellec S, Le Cesne A, Blay JY, Cousin P, Chaigneau L, Bompas E, Piperno-Neumann S, Bui-Nguyen B, Rios M, Delord JP, Penel N, Chevreau C. Efficacy of trabectedin in malignant solitary fibrous tumors: a retrospective analysis from the French Sarcoma Group. BMC Cancer. 2015 Oct 15;15:700. doi: 10.1186/s12885-015-1697-8. PMID 26472661
- [Background] Domont J, Massard C, Lassau N, Armand JP, Le Cesne A, Soria JC. Hemangiopericytoma and antiangiogenic therapy: clinical benefit of antiangiogenic therapy (sorafenib and sunitinib) in relapsed malignant haemangioperyctoma /solitary fibrous tumour. Invest New Drugs. 2010 Apr;28(2):199-202. doi: 10.1007/s10637-009-9249-1. Epub 2009 Apr 8. No abstract available. PMID 19352594
- [Background] Park MS, Patel SR, Ludwig JA, Trent JC, Conrad CA, Lazar AJ, Wang WL, Boonsirikamchai P, Choi H, Wang X, Benjamin RS, Araujo DM. Activity of temozolomide and bevacizumab in the treatment of locally advanced, recurrent, and metastatic hemangiopericytoma and malignant solitary fibrous tumor. Cancer. 2011 Nov 1;117(21):4939-47. doi: 10.1002/cncr.26098. Epub 2011 Apr 8. PMID 21480200
- [Background] Valentin T, Fournier C, Penel N, Bompas E, Chaigneau L, Isambert N, Chevreau C. Sorafenib in patients with progressive malignant solitary fibrous tumors: a subgroup analysis from a phase II study of the French Sarcoma Group (GSF/GETO). Invest New Drugs. 2013 Dec;31(6):1626-7. doi: 10.1007/s10637-013-0023-z. Epub 2013 Sep 5. PMID 24005614
- [Background] Stacchiotti S, Tortoreto M, Baldi GG, Grignani G, Toss A, Badalamenti G, Cominetti D, Morosi C, Dei Tos AP, Festinese F, Fumagalli E, Provenzano S, Gronchi A, Pennacchioli E, Negri T, Dagrada GP, Spagnuolo RD, Pilotti S, Casali PG, Zaffaroni N. Preclinical and clinical evidence of activity of pazopanib in solitary fibrous tumour. Eur J Cancer. 2014 Nov;50(17):3021-8. doi: 10.1016/j.ejca.2014.09.004. Epub 2014 Sep 27. PMID 25269954
- [Background] Martin-Broto J, Pousa AL, de Las Penas R, Garcia Del Muro X, Gutierrez A, Martinez-Trufero J, Cruz J, Alvarez R, Cubedo R, Redondo A, Maurel J, Carrasco JA, Lopez-Martin JA, Sala A, Meana JA, Ramos R, Martinez-Serra J, Lopez-Guerrero JA, Sevilla I, Balana C, Vaz A, De Juan A, Alemany R, Poveda A. Randomized Phase II Study of Trabectedin and Doxorubicin Compared With Doxorubicin Alone as First-Line Treatment in Patients With Advanced Soft Tissue Sarcomas: A Spanish Group for Research on Sarcoma Study. J Clin Oncol. 2016 Jul 1;34(19):2294-302. doi: 10.1200/JCO.2015.65.3329. Epub 2016 May 16. PMID 27185843